CLINICAL TRIAL: NCT00187603
Title: Protecting the 'Hood Against Tobacco: Cessation Project
Brief Title: Protecting the 'Hood Against Tobacco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Ruth Malone, Professor, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12AT-1700
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2005-08

CONDITIONS: Smoking
Keywords: tobacco; cessation; smoking; smoking cessation
MeSH Terms: conditions — Smoking; Smoking Cessation

INTERVENTIONS:
Behavioral: tobacco cessation program

SUMMARY:
Among all racial/ethnic groups, African Americans have the greatest risk of becoming ill or dying from tobacco-related diseases. Because of this disproportionate disease burden, it is particularly urgent that researchers focusing on tobacco control partner with African American communities. Intervention strategies which hold the tobacco industry accountable for its behavior are effective in changing views of tobacco use. In earlier work, the investigators found that information from internal tobacco industry documents, when shown to African American smokers, stimulated reflection about quitting and interest in disseminating information about industry targeting behaviors to others. However, to date there have been no attempts to utilize the information in industry documents as part of a smoking cessation intervention. In this project, the investigators will test whether a community co-developed, tailored quit-smoking program featuring exposures to African American-specific tobacco industry documents and media exercises in addition to proven individual quitting strategies can increase the number of people who quit smoking at six months and one year, as compared with usual care.

The specific aims of the project are to:

1. test, using statistics, how well an innovative community-based, culturally tailored quit-smoking program for African Americans works at 6 and 12 months;
2. test selected variables for how well they predict who will return to smoking;
3. use interviews to identify additional individual and/or community factors associated with successful quitting or relapse; and
4. collect information to evaluate the overall effectiveness of the CARA project collaborative efforts in developing and sustaining the project over time, enhancing community awareness of tobacco issues, and creation or enhancement of community tobacco control resources.

DETAILED DESCRIPTION:
Among all racial/ethnic groups, African Americans have the greatest risk of becoming ill or dying from tobacco-related diseases. Because of this disproportionate disease burden, it is particularly urgent that researchers focusing on tobacco control partner with African American communities. Intervention strategies which hold the tobacco industry accountable for its behavior are effective in changing views of tobacco use. In earlier work, we found that information from internal tobacco industry documents, when shown to African American smokers, stimulated reflection about quitting and interest in disseminating information about industry targeting behaviors to others. However, to date there have been no attempts to utilize the information in industry documents as part of a smoking cessation intervention. In this project, we will test whether a community co-developed, tailored quit-smoking program featuring exposures to African American-specific tobacco industry documents and media exercises in addition to proven individual quitting strategies can increase the number of people who quit smoking at six months and one year, as compared with usual care.

The specific aims of the project are to:

1. test, using statistics, how well an innovative community-based, culturally tailored quit-smoking program for African Americans works at 6 and 12 months;
2. test selected variables for how well they predict who will return to smoking;
3. use interviews to identify additional individual and/or community factors associated with successful quitting or relapse; and
4. collect information to evaluate the overall effectiveness of the CARA project collaborative efforts in developing and sustaining the project over time, enhancing community awareness of tobacco issues, and creation or enhancement of community tobacco control resources.

ELIGIBILITY:
Inclusion Criteria:

* African American adults who have used tobacco in the last month

Exclusion Criteria:

* Unable to read or speak English
* Dependence on other substances (except for marijuana)
* Disabling health conditions that would prevent participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Smoking cessation (cotinine validation) | at 6 and 12 months

SECONDARY OUTCOMES:
Qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Ruth E Malone, RN, PhD, Principal Investigator — Associate Professor UCSF
Locations (1):
- University of California San Francisco, San Francisco, California, United States